CLINICAL TRIAL: NCT01215721
Title: Vesicare™ (Solifenacin) in the Treatment of Urinary Incontinence After Radical Prostatectomy
Brief Title: Study to Determine Effects of Vesicare on Return to Continence Post - Radical Prostatectomy (Part II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Thomas E. Ahlering, Urology Account Contact, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-5720-2
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Results first posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2013-12

CONDITIONS: Urinary Incontinence
Keywords: Incontinence; Robotic Prostatectomy; Prostate Cancer
MeSH Terms: conditions — Urinary Incontinence; Prostatic Neoplasms | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vesicare (Experimental): Vesicare 5mg daily for 90 days was prescribed for men presenting with post-Robotic Assisted Radical Prostatectomy (RARP) severe incontinence.
  Interventions: Drug: Vesicare

INTERVENTIONS:
Drug: Vesicare — 5 mg daily
  Other Names: Vesicare (Solifenacin)

SUMMARY:
Prostate cancer is the most common non-cutaneous malignancy in men and is the 2nd leading cause of death from cancer in men. Radical prostatectomy is one of the treatment options available for organ-confined disease. Over 100,000 radical prostatectomies cases (total removal of the cancerous prostate by surgery) are performed in the United States yearly. Unfortunately nearly all of the men undergoing surgery report diminished Quality of Life (QOL) scores due in part due to a postoperative incontinence which may require the use of multiple urinary pads per day. Many of these men also report debilitating irritative voiding symptoms of urinary urgency and frequency, and have overall decreased urinary satisfaction scores. Abatement of these symptoms can take up to one year in men, and in 5-20% of patients symptoms may persist for longer periods.

Our recent published findings suggest that instability in the bladder muscle is likely an underlying etiology in postoperative urinary incontinence. This 'Detrusor Muscle' instability results in excess contractions of the urinary bladder ('urgency to urinate'), and can result in the feeling of needing to urinate more frequently. Consistent with this hypothesis of detrusor muscle instability, men with postoperative dribbling had more complaints with urgency, frequency and bother scores when queried with validated questionnaires. We suspect that a transient bladder muscle contraction may overcome the urinary sphincter valve resistance and result in the patient's dribbling of urine.

By treating the bladder muscle instability, we expect improved postoperative continence and improved quality of life in patients after undergoing surgery for total removal of a cancerous prostate. This pilot study will assess the statistical requirements for the number of subjects needed for a fully 'powered' randomized prospective study to fully evaluate whether medications such as solifenacin significantly improve patients' quality of urinary life and improve postoperative urinary incontinence after surgery.

*This study has been modified from the original protocol with the clinicaltrials.gov ID: NCT00581061.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have been diagnosed with prostate cancer and will undergo treatment for the disease as part of standard clinical care
* Patients that have multiple pad use a few days after standard of care catheter removal

Exclusion Criteria:

* Contra-indication to Solifenacin
* Narrow angle glaucoma
* Hepatic impairment
* Renal impairment
* CYP3A4 inhibitors (e.g. Ketoconazole)
* Gastric Retention (delayed or slow emptying of the stomach)
* Lives in a different country

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ahlering, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

REFERENCES:
- See also: Department of Urology | University of California, Irvine — http://www.urology.uci.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants are limited to men undergoing a robot assistered radical prostatectomy at the University of California, Irvine.
Pre-assignment Details: Only men who at the 6th or 7th day post-catheter removal are multiple pad users (3 pads or more) will be invited to participate in this trial.
Groups:
- Vesicare: Vesicare™ (Solifenacin) : 5 mg daily
Period: Overall Study
Arm/Group | Vesicare
Started | 40
Completed | 38
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Baseline Population: Men presenting with urinary incontinence requiring 3 pads or more at post-catheter day 6 or 7 after RARP (robotic assisted radical prostatectomy).
Arm/Group | Vesicare
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 40
Severely Incontinent Men Post RARP [Number; unit: Participants] — Only men who were experiencing severe incontinence were screened for possible enrollment on to the study. Men who were utilizing 3 or more pads at post-catheter day 6 or 7 were deemed severely incontinent, and were invited to participate int he trial.
  Participants | 40

OUTCOME MEASURES:

1. Primary Outcome: Time to Continence
Description: Days to zero pad continence were assessed by patient self-reported Pad free continence declaration card.
Time Frame: 12 months
Measure: Median (Standard Deviation); unit: Days to Continence
Groups:
- Vesicare, 5mg Treatment Group: Vesicare™ (Solifenacin) : 5 mg daily
Arm/Group | Vesicare, 5mg Treatment Group
Number analyzed (Participants) | 40
Days to Continence | 95 (128.8)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of 3 months from the time of medication administration.
Arm/Group | Vesicare, 5mg Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 2/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vesicare, 5mg Treatment Group (N=40)
Stomach Cramps (Gastrointestinal disorders) | 1 (1) — The patient was dehydrated while on the Vesicare medication, and as a result, suffered from a an episode of intense abdominal pain and constipation. The patient stopped taking the study medication and was not hospitalized.
Faintness, Flushing (General disorders) | 1 (1) — This patient was concomitantly taking the study medication Vesicare in addition to Viagra (Sildenafil citrate). During dinner the patient suffered shock, faintness, and flushing. The patient did visit the emergency room.

LIMITATIONS AND CAVEATS:
One limitation of this study was finding a reasonable Control group. This is problematic as symptoms that definitively identify detrusor overactivity preoperatively don't exist; hence we used pad usage 7 dys post catheter removal as a surrogate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No